CLINICAL TRIAL: NCT00566943
Title: Synovis Life Technologies, Inc., Peri-Strips Dry With Veritas Collagen Matrix Staple Line Reinforcement. The RESULTS Trial
Brief Title: Reinforcement of Surgical Staple Lines Using Peri-Strips Dry (PSD) With Veritas Collagen Matrix
Acronym: RESULTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP1007, Rev C
Record Dates: First submitted 2007-11-29; First posted 2007-12-04 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2011-07

CONDITIONS: Obesity
Keywords: Staple Line Reinforcement, Buttress
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients who have laparoscopic Roux-en-Y gastric by-pass surgery without staple line buttress material. No buttress material will be used on staple lines including stomach/pouch, anastomostic junctions, (gastrojejunostomy (GJ) gastric to intestine, or jejunojejunostomy (JJ) intestine to intestine). intestine or mesentery.
  Patients who have laparoscopic Roux-en-Y gastric by-pass surgery without buttress at the GJ anastomosis. Linear buttress at the stomach/pouch staple line is required.
  Interventions: Procedure: Roux-en-Y gastric by-pass surgery with no buttress
- PSD Veritas (Experimental): Linear Peri-Strips Dry Veritas Group: Patients who have laparoscopic Roux-en-Y gastric by-pass surgery with PSD Veritas used as a staple line buttress at the stomach/pouch.
  In addition to buttress of the stomach/pouch, patients may have PSD Veritas linear buttress at any of the following staple lines: intestine, mesentery, or anastomosis junction (gastrojejunostomy (GJ) gastric to intestine, or jejunojejunostomy (JJ) intestine to intestine).
  Circular Peri-Strips Dry Veritas Group: Patients who have laparoscopic Roux-en-Y gastric by-pass surgery with PSD Veritas circular buttress used as a staple line buttress at the GJ anastomosis. Linear buttress at the stomach/pouch is required.
  Interventions: Device: PSD Veritas Collagen Matrix

INTERVENTIONS:
Device: PSD Veritas Collagen Matrix — Roux-en-Y gastric by-pass surgery. Surgeon creates a small pouch from the stomach and then by-passes a large portion of the small intestine. The body cannot absorb as many calories or nutrients thus resulting in weight loss.
  Arms: PSD Veritas
Procedure: Roux-en-Y gastric by-pass surgery with no buttress — Patients who have laparoscopic Roux-en-Y gastric by-pass surgery without staple line buttress material. No buttress material will be used on staple line including stomach/pouch, anastomostic junctions, (gastrojejunostomy (GJ) gastric to intestine, or jejunojejunostomy (JJ) intestine to intestine intestine to mesentery.
  Arms: Control

SUMMARY:
The purpose of this study is to verify the performance of PSD Veritas to provide staple line protection during surgical procedures for obesity.

DETAILED DESCRIPTION:
The purpose of the study is to verify the performance of PSD Veritas in providing staple line protection for surgical procedures that buttress the stomach and other staple lines during roux-en-Y surgery. The study is designed as two separate patient groups. One will enroll patients into a group where linear staple lines are buttressed at the stomach. The second portion of the trial will enroll patients into a group where the circular staple line at the GJ and linear staple lines at the stomach are buttressed with PSD Veritas.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older
* Patient willing to comply with follow-up evaluations
* Patient understands nature of procedure and provides informed consent
* Female patient has stated that she is not pregnant and will not become pregnant during trial.

Exclusion Criteria:

* Patient currently enrolled in another device/drug trial that competes for same patient population
* Patient with short life expectancy (12 months) wherever the cause is not linked to obesity
* BMI is equal or less than 40 and equal to or less than 65
* Patient does not meet National Institute of Health (NIH) criteria for gastric by-pass surgery
* Patient has had previous buttress or other material used in the staple lines that will affect the outcome of this trial.
* Patient has known sensitivity to bovine material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger De La Torre, MD, Principal Investigator — Division of General Surgery University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at one surgical site in the US from approximately March 2006 through May 2008. One hundred one subjects were entered into the study.
Pre-assignment Details: Subjects were excluded from the study if their Body Mass Index was less than or equal to 35 or greater than or equal to 65. Subjects could not have a life expectancy of less than 12 months nor a known sensitivity to bovine material.
Groups:
- Control: control arm where no buttress is used on stomach or GJ anastomosis staple lines.
- PSD Veritas: PSD Veritas is used as a buttress for staple lines of the stomach and/or GJ anastomosis. Linear and circular refer to the shapes of the Veritas.
Period: Overall Study
Arm/Group | Control | PSD Veritas
Started | 52 | 49
Completed | 52 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PSD Veritas | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 49 | 101
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.93 (9.18) | 46.61 (10.2) | 45.3 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 40 | 87
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 52 | 49 | 101

OUTCOME MEASURES:

1. Primary Outcome: Linear and Circular Arm: Number of Subjects With Major Gastric Related Adverse Events Comparison Between Control and PSD Veritas Groups.
Description: Adverse events as measured through hospital discharge and 30 days post-discharge in both the linear and circular arms of the study.
Time Frame: Discharge/ 30 days Linear Discharge/30/90 days Circular
Measure: Number; unit: Participants
Groups:
- Number of Subjects in Control Group: control arm where no buttress is used on stomach or GJ anastomosis staple lines.
- Number of Subjects in PSD Veritas Group: PSD Veritas is used as a buttress for staple lines of the stomach and/or GJ anastomosis.
Arm/Group | Number of Subjects in Control Group | Number of Subjects in PSD Veritas Group
Number analyzed (Participants) | 52 | 49
Participants | 3 | 2

2. Primary Outcome: Linear and Circular Arm: Number of Participants With a Leak as Determined by a Comparison of Control Group to PSD Veritas Group.
Description: Leak as determined by a comparison of control group to PSD Veritas group in both linear and circular arms.
Time Frame: Discharge/30 Linear Discharge/30/90 days Circular
Measure: Number; unit: Participants
Arm/Group | Control | PSD Veritas
Number analyzed (Participants) | 52 | 49
Participants | 0 | 2

3. Secondary Outcome: Linear Arm: Comparison of Use of Endoclips or Sutures Used for Bleeding in Control Group Versus PSD Veritas Group
Description: Comparison of number of subjects who required use of Endoclips or sutures for bleeding in Control group versus the number of subjects who required use of Endoclips or sutures for bleeding in PSD Veritas group in the linear arm of the study.
Time Frame: Discharge and 30 days
Measure: Number; unit: Participants
Groups:
- Number of Subjects in Control Arm: control arm where no buttress is used on stomach or GJ anastomosis staple lines.
- Number of Subjects in PSD Veritas Arm Linear: PSD Veritas is used as a buttress for staple lines of the stomach and/or GJ anastomosis.
Arm/Group | Number of Subjects in Control Arm | Number of Subjects in PSD Veritas Arm Linear
Number analyzed (Participants) | 26 | 25
Participants | 10 | 6

4. Secondary Outcome: Number of Participants With Stricture Requiring Intervention Between Control Group and PSD Veritas Group. Bleeding Assessment of Control Group to PSD Veritas.
Description: Stricture requiring intervention comparison between control group and PSD Vertas group. Bleeding assessment comparison of control group to PSD Veritas Group. These results will combine both stricture and bleeding since this was how it was entered in to the database.
Time Frame: Discharge, 30 and 90 days
Measure: Number; unit: participants
Groups:
- Number of Subjects in PSD Veritas Arm: PSD Veritas is used as a buttress on stomach and/or GJ anastomosis.
Arm/Group | Number of Subjects in Control Arm | Number of Subjects in PSD Veritas Arm
Number analyzed (Participants) | 26 | 24
participants | 1 | 3

ADVERSE EVENTS:
Arm/Group | Control | PSD Veritas
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No